CLINICAL TRIAL: NCT06929403
Title: Effect of Dietary Supplement Containing Bergamot and Plant Sterols Extract on Serum Lipid Profile
Brief Title: Effect of Bergamot and Plant Sterols Extract on Serum Lipid Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Hande Seven Avuk, Assistant Professor, Head of Nutrition and Dietetic Department, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BERGAMIAPLANTSTEROLSTUDY
Record Dates: First submitted 2025-04-06; First posted 2025-04-16 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-04

CONDITIONS: Dyslipidemia; Cardiac Disease; Cardiovascular Diseases
Keywords: dyslipidemia; hyperlipidemia; plant sterols; Bergamot; complementary therapy
MeSH Terms: conditions — Dyslipidemias; Heart Diseases; Cardiovascular Diseases; Hyperlipidemias | interventions — Diet; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Diet Group (Active Comparator): Low-fat, low-cholesterol heart-protective diet
  Interventions: Behavioral: Diet
- Supplement Group (Experimental): Plant sterol/stanol supplement with bergamot
  Interventions: Dietary Supplement: Diet supplementation
- Diet and Supplement Group (Experimental): Plant sterol/stanol supplement with bergamot and Low-fat, low-cholesterol heart-protective diet
  Interventions: Behavioral: Diet; Dietary Supplement: Diet supplementation

INTERVENTIONS:
Behavioral: Diet — Low-fat, low-cholesterol heart-protective diet
  Other Names: Low-fat, low-cholesterol heart-protective diet
  Arms: Diet Group; Diet and Supplement Group
Dietary Supplement: Diet supplementation — 2 tablets/daily bergamot and plant sterol/stanol supplement (375 mg bergamot fruit extract, 800 mg plant sterols and 150 mg flavonoids) for 12 weeks
  Arms: Diet and Supplement Group; Supplement Group

SUMMARY:
The consumption of 2 grams of plant sterols per day has been demonstrated to positively affect total cholesterol and low density lipoprotein (LDL) cholesterol, as supported by various clinical guidelines. These compounds do not exhibit any adverse side effects. The European Society of Cardiology's Dyslipidemia Guidelines indicate that among lifestyle modifications aimed at reducing total cholesterol and LDL, the consumption of functional foods enriched with phytosterols should be included as a high-level recommendation.

Bergamot is a citrus fruit rich in flavonoids. Research on bergamot fruit extract has indicated its ability to lower total cholesterol, LDL cholesterol, and triglyceride levels while increasing high density lipoprotein(HDL) cholesterol levels. Furthermore, evidence suggests that it may help reduce high serum uric acid levels, which can pose a risk for cardiovascular diseases. The flavonoids in bergamot fruit extract contribute to the reduction of cholesterol synthesis in the liver. Additionally, it has a high capacity to prevent LDL oxidation. A study on individuals with metabolic syndrome observed significant and sustained reductions in serum cholesterol, triglyceride levels, and glucose in those consuming bergamot. This effect was accompanied by significant improvements in vascular reactivity in patients with hyperlipidemia and elevated serum glucose levels.

Bergamot also exhibits the ability to inhibit 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase. Due to their structural similarity to cholesterol, plant sterols help block the intestinal absorption of dietary cholesterol. They provide benefits at the absorption level and increase cholesterol excretion via bile and fecal pathways. The existence of known side effects associated with cholesterol-lowering medications, such as statins- including muscle cramps, myopathy, increased risk of muscle toxicity, liver damage, and neuropathy-has created a need for complementary or alternative approaches to treating dyslipidemia. This research will consider the potential of both plant sterols and bergamot as dietary supplements.

While cholesterol-lowering diets assist in reducing LDL, glucose, total cholesterol, and triglyceride levels, they do not enhance HDL levels. Because bergamot is known to increase HDL, it could provide an additional benefit in lipid profile regulation. A meta-analysis that studied various phytochemical supplements found that bergamot was the most effective in reducing total cholesterol, LDL, and triglyceride levels while increasing HDL levels. This study examines the effects of dietary supplementation containing plant sterols and bergamot on blood lipid profiles.

DETAILED DESCRIPTION:
This randomised clinical study, which aims to recruit 69 participants, will include individuals with abnormalities in their blood lipid profiles. Participants will be randomly assigned to one of three groups: Group 1 will receive a cholesterol-lowering diet; Group 2 will take bergamot with phytosterol/stanol supplements; and Group 3 will follow both a cholesterol-lowering diet and consume bergamot with phytosterol/stanol supplements. Participation in the study is voluntary and ethics committee approval has been obtained. Participants will take 2 tablets of bergamot and phytosterol/stanol supplements daily for 12 weeks, either on an empty stomach or with meals. Each 2-tablet dose will contain 375 mg of bergamot fruit extract containing 150 mg of flavonoids and 800 mg of plant sterols obtained from coniferous trees. Participants will be given detailed information about the study at the beginning and those who wish to participate will be asked to sign an informed consent form. Sample Size The sample size for the study was calculated using G*Power 3.1.9.7 software. Considering the research design, sample calculations were performed using ANOVA F test for group differences. Based on Cohen's medium effect size (d=0.5), 0.05 significance level (α=0.05) and desired power of 0.95, the minimum sample size required for inclusion in the study was determined as 66.

Statistical Analyses The findings of the study will be analyzed using Statistical Package for Social Sciences (IBM-SPSS) version 25. In the thesis, categorical variables will be summarized using frequency distributions, while quantitative variables will be defined using mean, standard deviation, minimum and maximum values. In order to reveal the relationships between variables and the differences between variable levels, both parametric and nonparametric methods will be used depending on the normality of the data. The normality of quantitative variables will be evaluated using Kolmogorov-Smirnov and Shapiro-Wilk tests. Parametric methods will be used for variables that show a normal distribution, and nonparametric alternatives will be used for variables that do not conform to a normal distribution. Significance will be determined at the p<0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Adults individuals who were diagnosed hyperlipidemia
* Individuals suitable for taking supplement

Exclusion Criteria:

* Chronic liver disease,
* Chronic kidney disease,
* Heart failure, infarction or cerebrovascular disease,
* Pregnant and breastfeeding women,
* Severe psychiatric disorders,
* Oncological diseases,
* People using medications that may interact with black seed oil (anticoagulant, antihypertensive, etc.)
* People using antilipidemic or anticholesterolemic medications in the last 3 months
* People with citrus allergies
* People who do not do heavy exercise
* People using any dietary supplements
* People with a known history of allergies
* People who do not regularly consume alcohol
* People with special dietary requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 61 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Biochemical Measurements - Fasting blood glucose | 12 weeks
  Fasting blood sugar (mg/dL) will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning and end of the study.
Biochemical Measurement - Lipid Profile | 12 weeks
  Participants' biochemical tests (total cholesterol, HDL cholesterol, LDL cholesterol, triglyceride, (mg/dL) will be analyzed in the hospital biochemistry laboratory using routine methods at the beginning and end of the study from blood samples taken by a nurse after at least 12 hours of fasting and without consuming alcohol for 24 hours before.
Biochemical Measurements - Liver Enzymes | 12 weeks
  Participants' liver enzymes tests (ALT and AST) (IU) will be analyzed in the hospital biochemistry laboratory using routine methods at the beginning and end of the study from blood samples taken by a nurse after at least 12 hours of fasting and without consuming alcohol for 24 hours before.
Biochemical Measurements - CRP | 12 weeks
  Participants' c-reactive protein tests (CRP) (mg/L) will be analyzed in the hospital biochemistry laboratory using routine methods at the beginning and end of the study from blood samples taken by a nurse after at least 12 hours of fasting and without consuming alcohol for 24 hours before.
Biochemical Measurements - Uric Acid Levels | 12 weeks
  Participants' serum uric acid tests (mg/dL) will be analyzed in the hospital biochemistry laboratory using routine methods at the beginning and end of the study from blood samples taken by a nurse after at least 12 hours of fasting and without consuming alcohol for 24 hours before.
Anthropometric Measurements - Body weight (kg) | 12 weeks
  At the beginning and end of the study, body weights (kg) will be measured using a bioelectrical impedance (BIA) device with a sensitivity of 50 grams in accordance with the measurement standards.
Anthropometric Measurements - Height | 1 week
  Height (cm) will be measured with a stadiometer in the Frankfort plane, standing and with the head upright.
Body Mass Index | 12 weeks
  The body mass index (BMI) of the participants will calculated according to the body weight (kg) / height (m)2 formula.
Body Mass Index Classification | 12 weeks
  The body mass index (BMI) of the participants is classified according to the World Health Organization (WHO) criteria. BMI ≤ 18.5 kg/m2 is underweight, between 18.5-24.99 kg/m2 is normal, ≥ 25 kg/m2 is overweight, and ≥ 30 kg/m2 is obese.
Anthropometric Measurements - Fat Mass | 12 weeks
  At the beginning and end of the study, body fat mass (kg) analysis will be performed using a bioelectrical impedance (BIA) device, paying attention to measurement standards.
Anthropometric Measurements - Fat ratio calculation | 12 weeks
  At the beginning and end of the study, body composition analyses will be performed using a bioelectrical impedance (BIA) device with measurement standards. According to the BIA analysis, fat percentage (%) will be calculated as the ratio of total body fat weight to total body weight.
Anthropometric Measurements - Fat-free mass | 12 weeks
  At the beginning and end of the study, fat-free mass (kg) will be analyzed using a bioelectrical impedance (BIA) device, paying attention to measurement standards.
Anthropometric Measurements - Muscle mass | 12 weeks
  At the beginning and end of the study, lean muscle mass (kg) will be analyzed using a bioelectrical impedance (BIA) device, paying attention to measurement standards.
Anthropometric Measurements - Total body water | 12 weeks
  At the beginning and end of the study, total body water (kg) will be analyzed using a bioelectrical impedance (BIA) device, paying attention to measurement standards.
Anthropometric Measurements - Waist circumference | 12 weeks
  At the beginning and end of the study, waist circumference will be measured with a non-flexible tape measure at the midpoint between the lowest rib and the crystalline prominence.
Anthropometric Measurements - Hip circumference | 12 weeks
  At the beginning and end of the study, the individual will be asked to stand upright with their arms at their sides and their feet side by side when measuring hip circumference. The Frankfort plane will be provided. The individual will be measured with a tape measure from the right side, determining the highest point of the hip (from the side).
Anthropometric Measurements - Waist/Height Ratio | 12 weeks
  Waist/height ratio will be obtained by dividing waist circumference by height at the beginning and end of the study.
Anthropometric Measurements - Waist/Hip Ratio | 12 weeks
  Waist/hip ratio will be obtained by dividing waist circumference by hip circumference.

SECONDARY OUTCOMES:
Physical Activity Levels | 1 week
  The International Physical Activity Questionnaire (IPAQ) Short Form, developed by Craig et al. and whose Turkish validity and reliability study was conducted by Öztürk, will be used to assess the physical activity levels of the participants. In the IPAQ short form (7 questions) assessment, the energy required for activities will be calculated with the Metabolic Equivalent Task minutes per week (MET-minutes) score. The calculation of the total score includes the sum of the duration (minutes) and frequency (days) of walking, moderate-intensity activity and vigorous activity. The physically inactive group is determined as those below 600 MET-min/week, moderately active between 600-3000 MET-min/week, active above 3000 MET-min/week, very active above 1500 MET-min/week and at least 3 days of vigorous activity or above 3000 MET-min/week and at least 7 days of walking.
Food Consumption Record | 3 days
  The food consumption record will be taken to evaluate the nutritional status of the participants. Food consumption records will be evaluated in the BeBIS (Nutrition Information System) program and the daily energy (kcal) intake will be calculated.
Food Consumption Record | 3 days
  The food consumption record will be taken to evaluate the nutritional status of the participants. Food consumption records will be evaluated in the BeBIS (Nutrition Information System) program and the daily carbohydrate (g), protein (g), fat (g), saturated fat (g), monounsaturated fatty acid (g), polyunsaturated fatty acid (g), omega-3 fatty acids (g), omega-6 fatty acids (g), and fiber (g) intake will be calculated.
Food Consumption Record | 3 days
  The food consumption record will be taken to evaluate the nutritional status of the participants. Food consumption records will be evaluated in the BeBIS (Nutrition Information System) program and the daily vitamin A (µg), vitamin D (µg), vitamin K (µg), folate (µg), and vitamin B12 (µg) intake will be calculated.
Food Consumption Record | 3 days
  The food consumption record will be taken to evaluate the nutritional status of the participants. Food consumption records will be evaluated in the BeBIS (Nutrition Information System) program and the daily vitamin E (mg), thiamine (mg), riboflavine (mg), niacin (mg), vitamine B5 (mg), vitamin B6 (mg), vitamin C, sodium (mg), potassium (mg), calcium (mg), magnesium (mg), phosphor (mg), iron (mg), zinc (mg), copper (mg), cholesterol (mg) intake will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Seven Avuk, Principal Investigator — İstanbul Bilgi University
Locations (1):
- İstanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norgan NG. Laboratory and field measurements of body composition. Public Health Nutr. 2005 Oct;8(7A):1108-22. doi: 10.1079/phn2005799. PMID 16277823
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Guasch-Ferre M, Babio N, Martinez-Gonzalez MA, Corella D, Ros E, Martin-Pelaez S, Estruch R, Aros F, Gomez-Gracia E, Fiol M, Santos-Lozano JM, Serra-Majem L, Bullo M, Toledo E, Barragan R, Fito M, Gea A, Salas-Salvado J; PREDIMED Study Investigators. Dietary fat intake and risk of cardiovascular disease and all-cause mortality in a population at high risk of cardiovascular disease. Am J Clin Nutr. 2015 Dec;102(6):1563-73. doi: 10.3945/ajcn.115.116046. Epub 2015 Nov 11. PMID 26561617
- [Background] Osadnik T, Golawski M, Lewandowski P, Morze J, Osadnik K, Pawlas N, Lejawa M, Jakubiak GK, Mazur A, Schwingschackl L, Gasior M, Banach M. A network meta-analysis on the comparative effect of nutraceuticals on lipid profile in adults. Pharmacol Res. 2022 Sep;183:106402. doi: 10.1016/j.phrs.2022.106402. Epub 2022 Aug 18. PMID 35988871
- [Background] Racette SB, Lin X, Lefevre M, Spearie CA, Most MM, Ma L, Ostlund RE Jr. Dose effects of dietary phytosterols on cholesterol metabolism: a controlled feeding study. Am J Clin Nutr. 2010 Jan;91(1):32-8. doi: 10.3945/ajcn.2009.28070. Epub 2009 Nov 4. PMID 19889819
- [Background] Ferro Y, Maurotti S, Mazza E, Pujia R, Sciacqua A, Musolino V, Mollace V, Pujia A, Montalcini T. Citrus Bergamia and Cynara Cardunculus Reduce Serum Uric Acid in Individuals with Non-Alcoholic Fatty Liver Disease. Medicina (Kaunas). 2022 Nov 26;58(12):1728. doi: 10.3390/medicina58121728. PMID 36556930
- [Background] Gliozzi M, Walker R, Muscoli S, Vitale C, Gratteri S, Carresi C, Musolino V, Russo V, Janda E, Ragusa S, Aloe A, Palma E, Muscoli C, Romeo F, Mollace V. Bergamot polyphenolic fraction enhances rosuvastatin-induced effect on LDL-cholesterol, LOX-1 expression and protein kinase B phosphorylation in patients with hyperlipidemia. Int J Cardiol. 2013 Dec 10;170(2):140-5. doi: 10.1016/j.ijcard.2013.08.125. Epub 2013 Sep 8. PMID 24239156
- [Background] Toth PP, Patti AM, Nikolic D, Giglio RV, Castellino G, Biancucci T, Geraci F, David S, Montalto G, Rizvi A, Rizzo M. Bergamot Reduces Plasma Lipids, Atherogenic Small Dense LDL, and Subclinical Atherosclerosis in Subjects with Moderate Hypercholesterolemia: A 6 Months Prospective Study. Front Pharmacol. 2016 Jan 6;6:299. doi: 10.3389/fphar.2015.00299. eCollection 2015. PMID 26779019
- [Background] Gylling H, Plat J, Turley S, Ginsberg HN, Ellegard L, Jessup W, Jones PJ, Lutjohann D, Maerz W, Masana L, Silbernagel G, Staels B, Boren J, Catapano AL, De Backer G, Deanfield J, Descamps OS, Kovanen PT, Riccardi G, Tokgozoglu L, Chapman MJ; European Atherosclerosis Society Consensus Panel on Phytosterols. Plant sterols and plant stanols in the management of dyslipidaemia and prevention of cardiovascular disease. Atherosclerosis. 2014 Feb;232(2):346-60. doi: 10.1016/j.atherosclerosis.2013.11.043. Epub 2013 Nov 23. PMID 24468148
- [Background] Catapano AL, Graham I, De Backer G, Wiklund O, Chapman MJ, Drexel H, Hoes AW, Jennings CS, Landmesser U, Pedersen TR, Reiner Z, Riccardi G, Taskinen MR, Tokgozoglu L, Verschuren WMM, Vlachopoulos C, Wood DA, Zamorano JL, Cooney MT; ESC Scientific Document Group. 2016 ESC/EAS Guidelines for the Management of Dyslipidaemias. Eur Heart J. 2016 Oct 14;37(39):2999-3058. doi: 10.1093/eurheartj/ehw272. Epub 2016 Aug 27. No abstract available. PMID 27567407
- [Background] Expert Dyslipidemia Panel of the International Atherosclerosis Society Panel members. An International Atherosclerosis Society Position Paper: global recommendations for the management of dyslipidemia--full report. J Clin Lipidol. 2014 Jan-Feb;8(1):29-60. doi: 10.1016/j.jacl.2013.12.005. Epub 2013 Dec 17. PMID 24528685